CLINICAL TRIAL: NCT02870348
Title: A Multi-Center, Open-Label Study to Evaluate the Long-term Safety of Weekly Intravenous Infusions of Alpha1-Proteinase Inhibitor (Human) in Japanese Subjects With Alpha1 Antitrypsin Deficiency
Brief Title: Long-term Safety of Alpha1-Proteinase Inhibitor (Human) in Japanese Subjects With Alpha1 Antitrypsin Deficiency (GTI1401-OLE)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Grifols Japan K.K. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI1401-OLE; JapicCTI-163194 (Other: JapicCTI)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Results first posted 2022-03-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Alpha1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — Mp alpha1 receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpha-1 MP (Experimental): Participants received IV infusion of 60 mg/kg Alpha-1 MP administered weekly for mean duration of 213 weeks.
  Interventions: Biological: Alpha-1 MP

INTERVENTIONS:
Biological: Alpha-1 MP — Alpha-1 MP is a stable, sterile, lyophilized preparation of human alpha1-PI, also known as alpha1-antitrypsin.
  Other Names: Prolastin-C

SUMMARY:
This is a multi-center, open-label study to evaluate the long-term safety of weekly intravenous (IV) infusions of 60 mg/kg alpha1-PI (human), modified process (Alpha-1 MP) in adult participants with Alpha1 Antitrypsin Deficiency (AATD) in Japan who have completed Study GTI1401 (NCT02870309).

DETAILED DESCRIPTION:
This is a multi-center, open-label study to evaluate the long-term safety of weekly IV infusions of 60 mg/kg Alpha-1 MP in adult participants with AATD in Japan who have completed Study GTI1401. Study GTI1401 is being conducted to evaluate the safety and pharmacokinetics (PK) of Alpha-1 MP in participants with AATD in Japan. In the current study, GTI1401-OLE, participants will be administered 60 mg/kg Alpha-1 MP by weekly IV infusion for approximately 1 year (can be renewed annually with the consent of the participants unless the sponsor informs of discontinuation of this OLE trial) to assess the long-term safety of Alpha-1 MP in participants with AATD. This study will be conducted at up to 5 centers in Japan.

At the Week 9 Visit of Study GTI1401, after giving consent, on the same day, participants will be assessed for eligibility at Screening/Extension (Ext) Week 1 Visit for this extension study, Study GTI1401-OLE. If eligible, participants will be administered weekly IV infusions of 60 mg/kg Alpha-1 MP for approximately 1 year or longer. The Week 9 Visit of GTI1401 will be the End of Study Visit for the participants who are enrolled in Study GTI1401-OLE.

Participants in Study GTI1401-OLE will have the option to remain in Study GTI1401-OLE and continue to receive weekly IV infusions of 60 mg/kg Alpha-1 MP for another year or longer. If participants plan to conclude their participation in the study (GTI1401-OLE) early (before Ext. Week 52), participants will be asked to complete the End of Study Follow-Up Assessments, which will be scheduled 4 weeks after the last infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who complete participation in Study GTI1401 (i.e., have completed the study through the Week 9 Visit).
* Subjects who will and are able to provide written informed consent.

Exclusion Criteria:

* Subjects with newly diagnosed severe concomitant disease including, but not limited to, congestive heart failure and liver cirrhosis.
* Subjects with newly diagnosed malignant tumor (including malignant melanoma; however, other forms of skin cancer are allowed).
* Female subjects who are pregnant, breastfeeding or, if of child-bearing potential, unwilling to practice a highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or abstinence) throughout the study or male subjects who have a partner who is of child-bearing potential and is unwilling to practice a highly effective method of contraception throughout the study.
* Subjects with clinical signs and symptoms of active hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) viral infection at the Week 9 Visit of Study GTI1401 and viral infection is further confirmed by testing.
* Subjects with current evidence of smoking or has a positive urine cotinine test at the Week 9 Visit in Study GTI1401 that is due to smoking.
* Subjects who currently participate in a study of another investigational product (other than Alpha-1 MP).
* Subjects who have difficulty in adhering to the protocol or its procedures, in the opinion of the investigator.
* Subjects who have medical conditions that may confound the results of this clinical trial or may endanger these subjects during their participation in this clinical trial in the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Hiroskai University Hospital, Aomori
  - Hokkaido University Hospital, Hokkaido
  - Juntendo University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seyama K, Suzuki M, Tasaka S, Nukiwa T, Sato T, Konno S, Sorrells S, Chen J, Aragones ME, Minamino H. Long-term safety of Prolastin(R)-C, an alpha1-proteinase inhibitor, in Japanese patients with alpha1-antitrypsin deficiency. Respir Investig. 2022 Nov;60(6):831-839. doi: 10.1016/j.resinv.2022.07.001. Epub 2022 Aug 12. PMID 35970714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 investigative sites in Japan from 29 July 2016 to 16 February 2021.
Pre-assignment Details: Participants with diagnosis of alpha1-antitrypsin deficiency (AATD) who completed the Study GTI1401 (NCT02870309) were eligible to enroll in this open-label extension study. The Screening / Extension (Ext) Week 1 Visit and initiation of treatment for the current study (GTI1401-OLE) occurred on the same day as the Week 9 Visit of GTI1401 only for those participants who gave the consent for participation in the Study GTI1401-OLE.
Period: Overall Study
Arm/Group | Alpha-1 MP
Started | 4
Completed | 0
Not Completed | 4
Not completed — Participants were discontinued and assessed for entry into post-marketing study (GTI1401-EXP) | 4

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product or study treatment and which did not necessarily have a causal relationship with this administration. TEAEs were defined as any AE occurring after or on the first Alpha-1 MP infusion until the final visit of study.
Time Frame: From start of study drug administration through 30 days after last study drug infusion (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Number of Participants With Adverse Drug Reaction (ADRs)
Description: ADRs were defined as all noxious and unintended responses to a medicinal product or study treatment related to any dose. An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product or study treatment and which did not necessarily have a causal relationship with this administration.
Time Frame: From start of study drug administration through 30 days after last study drug infusion (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 2

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was considered serious in any of the following outcomes or deemed significant for any other reason: death; life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; congenital anomaly/birth defect.
Time Frame: From start of study drug administration through 30 days after last study drug infusion (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 2

4. Primary Outcome: Number of Participants With Discontinuations Due to Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product or study treatment and which did not necessarily have a causal relationship with this administration. An AE was considered serious in any of the following outcomes or deemed significant for any other reason: death; life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; congenital anomaly/birth defect.
Time Frame: From start of study drug administration through 30 days after last study drug infusion (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

5. Primary Outcome: Number of Participants With Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: COPD exacerbation was defined as an increase in respiratory symptoms (dyspnea, increased cough, and/or production of sputum) over baseline that usually requires medical intervention.
Time Frame: From start of study drug administration through 30 days after last study drug infusion (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs
Description: Vital signs included analysis of heart rate, blood pressure, respiratory rate, and temperature. Clinically significant findings in vital signs were based on investigator's discretion.
Time Frame: From start of study drug administration through 30 days after last study drug infusion (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Significant Findings in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included analysis of hematology, blood chemistry, and urinalysis. Clinically significant findings in clinical laboratory parameters were based on investigator's discretion.
Time Frame: Extension (Ext) Weeks 26, 52, 78, 104, 130, 156,182, 208 (prior to study drug administration) until end of study (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

8. Primary Outcome: Number of Participants With Clinically Significant Findings in Pulmonary Function Tests (PFTs)
Description: Pulmonary function tests were measured by spirometry. It included Forced Expired Volume in 1 second (FEV1), Forced Vital Capacity (FVC), which were performed according to American Thoracic Society/ European Respiratory Society (ATS/ERS) guidelines. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. PFTs were performed before infusion both pre- and post-bronchodilator administration. The post-bronchodilator PFT was performed 15 to 30 minutes after bronchodilator administration. The same bronchodilator was used throughout the study. Clinically significant findings in pulmonary function tests were based on investigator's discretion.
Time Frame: as for outcome 7
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

9. Primary Outcome: Trough Levels of Alpha1- Proteinase Inhibitor
Description: Alpha1-PI level was measured by nephelometry.
Time Frame: Extension (Ext) Weeks 12, 24, 36, 48, 64, 76, 88, 100, 116, 128, 140, 152, 168, 180, 192, 204 (prior to study drug administration) until end of study (Up to 228 weeks)
Population: Safety Population included all participants who received any amount of Alpha-1 MP.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
milligram/deciliter (mg/dL) | 55.734 (4.9928)

ADVERSE EVENTS:
Time Frame: From start of study drug administration through 30 days after last study drug infusion (Up to 228 weeks)
Description: Safety Population included all participants who received any amount of Alpha-1 MP.
Arm/Group | Alpha-1 MP
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha-1 MP (N=4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha-1 MP (N=4)
Arrhythmia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Eyelid pain (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 1
Influenza virus test positive (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT02870348/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT02870348/SAP_001.pdf